CLINICAL TRIAL: NCT01297530
Title: An Open-label, Phase I, Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY87-2243 Given Once Daily in Subjects With Advanced Malignancies
Brief Title: Clinical Study to Evaluate the Maximum Tolerated Dose of BAY87-2243 in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head of Clinical Sciences, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15044; 2010-023403-10 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Neoplasms
Keywords: Phase I; Dose Escalation; Hypoxia inducible factor 1 alpha; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — 1-cyclopropyl-4-(4-((5-methyl-3-(3-(4-(trifluoromethoxy)phenyl)-1,2,4-oxadiazol-5-yl)-1H-pyrazol-1-yl)methyl)pyridin-2-yl)piperazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY87-2243

INTERVENTIONS:
Drug: BAY87-2243 — Oral administration once daily in a continuous schedule. Starting dose will be 5 mg and dose will be escalated dependent on any dose limiting toxicities.

SUMMARY:
This is the first study of this drug in human beings. Every patient will receive the drug, there is no placebo group. Patients with advanced tumors will be treated. Different groups of patients will receive different dosages to determine the safety and maximum tolerated dose (MTD) of BAY87-2243. The study will also assess how the drug is metabolized by the body, its biologic effects in the body, and changes in tumor size.

BAY87-2243 will be given as a tablet which dissolves in the gut. Based on findings from this study it may be later given as a tablet which dissolves in the stomach.

BAY87-2243 will be given per mouth, once a day, every day. Treatment will stop if the tumor continues to grow, if side effects occur which the patient can not tolerate or if the patients decides to exit treatment.

The study will be conducted in 3 - 4 centers in 3 countries (Norway, United Kingdom and Germany). The study will have a part where doses are escalated in different groups of patients. Each dose level will be evaluated in a new group of 3 - 6 subjects. This will be followed by an extension part where patients are treated at the highest tolerable dose in groups of up to 25 patients. The extension part will be described in an amendment to the study protocol later. The number of subjects estimated for this study will depend on the number of groups enrolled. The starting dose will be 5 mg given orally as a tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >/= 18 years
* Subjects with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and / or if in the judgement of the investigator, experimental treatment is clinically and ethically acceptable
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Life expectancy of at least 3 month
* Adequate bone marrow, liver, and renal functions

Exclusion Criteria:

* History of cardiac disease including congestive heart failure > NYHA (New York Heart Association) II, unstable angina (anginal symptoms at rest), or new-onset angina (within the past 3 months) or myocardial infarction within the past 6 months and cardiac arrhythmias requiring anti-arrhythmic therapy except for beta-blockers and digoxin
* History of ischemic cardiovascular disease
* Family history of long QT syndrome
* Persistent hypokalemia < 3.5 mmol/L
* History of cerebral ischemia including transient ischemic attack (TIA), prolonged reversible ischemic neurologic deficit (PRIND), and ischemic stroke within the past 6 months
* Known alcohol abuse
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C
* Diabetes mellitus treated with oral antidiabetics or insulin
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Active clinically serious infections of CTCAE > Grade 2 (Common Terminology Criteria for Adverse Events v4.02)
* Symptomatic metastatic brain or meningeal tumors unless the subject is > 6 months from definitive therapy, has no evidence of tumor growth on an imaging study within 4 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry.
* Unresolved specific chronic toxicity CTCAE > Grade 2
* Subjects may not receive potent inducers of CYP3A4, such as phenytoin, carbamazepine, and rifampicin, as the oral clearance of ondansetron may increase and ondansetron plasma concentrations may decrease due to antiemetic regimen
* Concomitant medication with metformin
* Concomitant medication with drugs known to prolong the QT interval
* Relevant pathological changes in the ECG such as a second or third-degree AV block, prolongation of the QRS complex over 120 ms or of the QT / QTc-interval over 450 ms in men and women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | Up to 3 years or longer if indicated
Maximum tolerated dose, measured by adverse event profile | Up to 3 years or longer if indicated

SECONDARY OUTCOMES:
Plasma concentrations of BAY87-2243, measured by Cmax, tmax, AUC(0-tn), AUC and half-life | Up to 3 years or longer if indicated
Biomarkers evaluation (analysis of carbonic anhydrase 9 and VEGF in plasma) | Up to 3 years or longer if indicated
Tumor response evaluation based on RECIST 1.1 every 2 cycles | Up to 3 years or longer if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Oslo, Norway
- Sutton, Surrey, United Kingdom